CLINICAL TRIAL: NCT02435953
Title: Transarterial Chemoembolization Plus Radiofrequency Ablation Versus Transarterial Chemoembolization Alone for Intermediate-stage Hepatocellular Carcinoma
Brief Title: TACE+RFA Versus TACE Alone for Intermediate-stage Hepatocellular Carcinoma
Acronym: TORCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ming Zhao (Other)
Responsible Party: Sponsor-Investigator, Ming Zhao, Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-FXY-089
Record Dates: First submitted 2015-05-03; First posted 2015-05-06 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Chemoembolization, Therapeutic; Ablation Techniques, RFA
Keywords: Hepatocellular Carcinoma,TACE,Chemoembolization, RFA,Intermediate-stage
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE-RFA (Experimental): RFA follows TACE when achieving ablation eligibility criteria defined in this study, with no more than four sessions of TACE.
  Interventions: Procedure: TACE; Procedure: RFA
- TACE alone (Active Comparator): On-demand TACE.
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — A catheter (or a microcatheter for cases where small vessels and branches cannot be accessed with a standard angiographic catheter) will be advanced selectively or superselectively into the right or left hepatic artery or the feeding arteries directly supplying the tumor. Depending on tumor size, location, blood supply, and liver function, the interventional radiologist administers a cytotoxic agent and lipiodol emulsion (30 mg lobaplatin, 30 mg pirarubicin, and < 15 mL lipiodol) through the catheter. Following drug infusion, embolization of the tumor vessels will be routinely performed using gelatin sponge particles.
Procedure: RFA — Commercial electrode systems are used and the ablation therapy is to be performed according to manufacturer's standard recommendations. All lesions are targeted with CT images during the RFA procedure.
  Arms: TACE-RFA

SUMMARY:
The current standard treatment for intermediate-stage HCC (BCLC stage B) is transcatheter arterial chemoembolization (TACE) alone. The combination of TACE with RFA has also reported to be an effective treatment for HCC. Some prospective studies have shown that TACE combined with RFA have better efficacy than any of them alone for early stage HCC (single tumor ≤5 cm). However, to the investigators' knowledge, there have not been any prospective studies to assess whether TACE combined sequentially with RFA is more effective than TACE alone for the treatment of intermediate-stage HCC. The investigators hypothesized that the combination of TACE and RFA might result in better patient survival than TACE alone. Thus, the purpose of this study was to prospectively compare the effects of sequential TACE-RFA with TACE alone for the treatment of intermediate-stage HCC. Intermediate-stage HCC in this study was defined as 2-3 intrahepatic lessions, largest tumor size 3-7 cm or 4-10 intrahepatic lessions, largest tumor size ≤7 cm; ECOG-PS 0; Child-pugh A or B7; no tumor thrombus or extrahepatic metastases.

ELIGIBILITY:
Inclusion Criteria:

* Multiple HCC (2-3 lesions), largest lesion 3-7 cm in diameter, or multiple HCC (4-10 lesions), each ≤ 7 cm in diameter
* No vascular invasion or etrahepatic metastases
* Eastern Cooperative Oncology Group Performance Status 0
* Child-Pugh Stage A or B7
* Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to procedure:

I.Adequate hematologic function:

1. WBC ≥ 4.0 x 109/L (stable, off any growth factor within 4 weeks of study drug administration)
2. Neutrophils ≥ 1.5 x 109/L (stable, off any growth factor within 4 weeks of study drug administration)
3. Platelets ≥ 60 x 109/L (transfusion to achieve this level is not permitted)
4. Hemoglobin ≥ 100 g/L (may be transfused to meet this requirement)

II.Adequate hepatic function:

1. Serum Aspartate Aminotransferase (AST) ≤ 5×ULN
2. Serum Alanine Aminotransferase (ALT) ≤ 5×ULN
3. Serum total bilirubin ≤ 51.3 μmol/L
4. Serum albumin ≥ 2.8 g/dL

III.Adequate coagulation function:

a)prothrombin activity ≥ 40%

IV.Adequate renal function:

a)Serum creatinine < 110 μmol/L

Exclusion Criteria:

* Previous local therapy completed less than 4 weeks prior to the dosing and, if present any related acute toxicity > grade 1
* Any contraindications for TACE/RFA procedure:

I.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 40%) II.Renal failure / insufficiency requiring hemodialysis or peritoneal dialysis. III.Known severe atheromatosis IV.Known uncontrolled blood hypertension (> 160/100 mmHg) V.Patients with known active bleeding (e.g. from GI ulcers, esophageal varices) within 2 months prior to baseline/screening visit or with history or evidence of inherited bleeding diathesis or coagulopathy VI.Clinically significant third space fluid accumulation (i.e., ascites requiring tapping despite use of diuretic or pleural effusion that either required tapping or is associated with shortness of breath)

* Evidence of hepatic discompensation (i.e., refractory ascites, esophageal or gastric variceal bleeding, or hepatic encephalophathy)
* Patients with any other malignancies within the last 3 years before study start
* History of HCC tumor rupture
* Clinically significant (CTC grade 3 or 4) venous or arterial thrombotic disease within past 6 months
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within past 6 months prior to study treatment
* Pregnant women or lactating women
* Be allergic to pirarubicin, lobaplatin and iodized oil

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2025-10 (Actual); Study Completion 2025-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (PFS-R) | From the date of randomization to the date of occurrence of radiologic disease progression as determined according to the RECIST v1.1, or death (by any cause), whichever occurs first, assessed up to 8 months.

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death (due to any cause), assessed up to 2.5 years.
Progression-free survival (PFS) according to HCC modified RECIST (PFS-m) | From the date of randomization to the date of occurrence of radiologic disease progression as determined according to the HCC modified RECIST, or death (by any cause), whichever occurs first, assessed up to 8 months.
unAblation-TACEable or unTACEable progression-free survival (uAT-PFS) | From the date of randomization to the date of the following untreatable progression or death by any cause, assessed up to 24 months.
Objective response rate (ORR) according to RECIST v1.1 (ORR-R) | From date of randomization until the date of study completion, an average of 8 months.
Objective response rate (ORR) according to mRECIST (ORR-m) | From date of randomization until the date of study completion, an average of 8 months.
Disease control rate (DCR) according to RECIST v1.1 (DCR-R) | From date of randomization until the date of study completion, an average of 8 months.
Disease control rate (DCR) according to mRECIST (DCR-m) | From date of randomization until the date of study completion, an average of 8 months.
Adverse Events | From enrollment to until 30 days following discontinuation of study treatment or until the initiation of the first subsequent therapy following discontinuation of study treatment (whichever occurs first).

OTHER OUTCOMES:
Time to advanced-stage (TTAS) | From randomization to disease progression to Barcelona Clinic Liver Cancer stage C (BCLC-C), assessed up to 2 years.
Time to extrahepatic spread (TTEHS) | From randomization to occurrence of extrahepatic metastasis, assessed up to 2 years.
Time to macrovascular invasion (TTMVI) | From randomization to occurrence of macrovascular invasion, assessed up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, doctor, Principal Investigator — Principal Investigator, Clinical Professor
Locations (1):
- Minimally Invasive Interventional Division, Medical Imaging Center, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China